CLINICAL TRIAL: NCT03665363
Title: Efficacy and Effectiveness of SCOPE for Intellectually Able Youths With Autism Spectrum Disorder- a Randomized Controlled Study
Brief Title: Evaluating the Efficacy and Effectiveness of SCOPE - RCT
Acronym: SCOPERCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Stiftelsen Promobilia (Unknown); Stiftelsen Sunnerdahls Handikappfond (Other); Stiftelsen Sven Jerrings fond (Unknown); L.J. Boëthius stiftelse (Unknown); Stiftelsen Frimurarna Barnhuset (Unknown); Stockholm County Council ALF/PPG (Unknown)
Responsible Party: Principal Investigator, Tatja Hirvikoski, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: SCOPERCT
Record Dates: First submitted 2018-09-03; First posted 2018-09-11 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Autism Spectrum Disorder; Transition
Keywords: Young adults; Psychoeducation; Internet-based intervention; Adolescents
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SCOPE (Experimental): Participants allocated to SCOPE, will receive an internet-based psychoeducation intervention, eight weeks of ASD-theme modules with coaching.
  Interventions: Other: SCOPE
- Self-study (Active Comparator): Participants allocated to self-study will receive eight weekly emails containing informative and relevant websites about ASD. The emails are accessed on the same platform as the experimental condition (SCOPE), no active contact with the coaches is available.
  Interventions: Other: Self-study
- Wait-list controls/Treatment as usual (No Intervention): Participants allocated to wait-list will receive prompts to answer outcome measures but otherwise no other contact with the study coordinators or coaches. Participants may receive treatment as usual.

INTERVENTIONS:
Other: SCOPE — SCOPE is a internet-delivered, coach-guided, psychoeducational intervention, intended to serve as a first-line intervention for intellectually able adolescents and young adults with ASD. The SCOPE program is based on information comprising neuropsychology, pedagogy, and also interdisciplinary clinical experience regarding ASD. The content is aimed at providing information about typical and specific impairments of ASD, as well as the associated strengths.
  Arms: SCOPE
Other: Self-study — Active control consisting of directed self-studies on internet.
  Arms: Self-study

SUMMARY:
The study will entail an evaluation of the feasibility, acceptability, efficacy and effectiveness of SCOPE coach supported internet-delivered psychoeducative program using a randomized controlled design in a clinical health care context.

An estimated n=175 will be needed to enable block randomisation according a 2:1:1 ratio to: 1) SCOPE internet-based psychoeducation intervention, 2) Self-study controls, who receive eight weekly emails containing informative and relevant websites about Autism Spectrum Disorder (ASD), 3) Wait-list controls.

DETAILED DESCRIPTION:
The internet-delivered intervention SCOPE was developed using a participatory research approach, i.e. in cooperation with the target group. SCOPE has eight ASD theme modules and weekly contact with an experienced clinician (coach) via a message function within the Swedish national platform for internet-delivered treatment (1177.se e-services).

The three treatment arms means that the self-study controls as well as the wait-list controls will have the option to take part of SCOPE the following semester after having completed the data collection process. The assessment of eligibility is conducted on the national platform for internet-delivered interventions using a web camera application or phone interview. The intake assessment covers depression symptoms and suicidality using MADRS-R, functional impairment using WHODAS 2.0 (WHO), and validation of autism core symptoms using OSU Autism and Social Responsiveness Scale.

Treatment expectancy and satisfaction will be measured using the Treatment Credibility Scale (see outcome measures) and an evaluation of each module.The criteria for feasibility were (1) attrition should be less than 40% and (2) the participants should attend at least 75% of the sessions. Efficacy-related measures will be gained through the primary outcome of improved knowledge about ASD. Secondary outcomes are mental health: symptoms of anxiety and depression; acceptance of diagnosis; and quality of life. In addition, measures of treatment credibility are also completed by the coaches. The measures will be analysed using a series of repeated measures ANOVAs (rmANOVAs) to analyse differences between treatment arms.

The recommended first-line intervention for ASD is psychoeducation. Psychoeducational interventions for transition-aged autistic youth have a very limited evidence base. Therefore, the effect of psychoeducation for the target group is difficult to discern, the current study would contribute significantly to the research field. The findings will be important especially as psychoeducation is a clinically common intervention, provided in a non-standardized way and without sufficient information of its effects.

Recruitment commenced during the autumn of 2016 and was completed in december 2020. Final n=144.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed autism spectrum disorder with IQ in the average range (>70) (diagnosed in accordance with the DSM or ICD-10 diagnostic manuals)
* relevant age group (16 to 25 years)
* active participation in the eight-week program
* sufficient Swedish language proficiency
* ability to log on and utilize an internet-based platform

Exclusion Criteria:

* current substance misuse (including the past three months)
* suicidal ideation,
* diagnosed with intellectual disability (according to DSM or ICD),
* diagnosed with traumatic brain injury (e.g., stroke),
* other severe psychiatric disorders (e.g., psychosis) or adverse psychosocial circumstances (e.g., being homeless) that would render participation unlikely or impossible.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Both biological sex or self-described gender identity will be registered.
Enrollment: 144 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Change in scores on the ASD Knowledge Quiz | Change in knowledge measured at baseline, immediately after the intervention and at three month follow-up
  16 questions about general knowledge about ASD. The questions are based on the eight modules in the interventions.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | Measured at baseline, immediately after the intervention and at three month follow-up
  Has 14 items scored 0 ("Often" ) - 3 ("Seldom"), subsequently summarized for an overall score; high scores indicate higher levels of depression or anxiety.
Acceptance and Action Questionnaire (AAQ-II) | Measured at baseline, immediately after the intervention and at three month follow-up
  Acceptance of the diagnosis was estimated, using a modified version of the AAQ-II. The current version focuses on acceptance of having an ASD diagnosis, using a seven-item scale ranging from 1 ("Never") to 7 ("Always"), and was then summarized for an overall score; high scores indicate low acceptance of the diagnosis. The item wording after adjustment to the current study were: (1) "My diagnosis makes it difficult for me to lead a life I could value"; (2) "I am afraid of my diagnosis"; (3) "I worry about not being able to control my worries and my feelings regarding my diagnosis"; (4) "My diagnosis prevents me from leading a fulfilling life"; (5) "My diagnosis creates problems in my life"; (6) "I feel uncomfortable with my diagnosis"; (7) "My diagnosis gets in the way of my success".
Brunnsviken Brief Quality of Life Inventory (BBQ) | Measured at baseline, immediately after the intervention and at three month follow-up
  A measure estimating quality of life using 12 items: using a scale ranging from 1 ("Not at all") to 4 ("Very much"), subsequently summarized for an overall score; high scores indicate high satisfaction with life.

OTHER OUTCOMES:
The Treatment Credibility Scale (TCS) | Measured at baseline, immediately after the intervention and at three month follow-up
  As a measure of feasibility TCS is used to measure the expectation of improvement and treatment credibility. The TCS is a visual analogue scale rated from "Low credibility"/ "Not at all" (0) to "High credibility"/"Very much" (10) and the score calculated is a mean of all items. The TCS was administered after providing thorough information and presentation of the treatment content at baseline and after completion of the treatment. The item wording after adjustment to the current study were: (1) How logical does SCOPE seem to you?; (2) How confident are you that you will learn more about autism from SCOPE?; (3) Would you recommend SCOPE to a friend with ASD?; (4) How successful do you feel this type of program would be in teaching about other diagnoses?; (5) How much do you think you will have learned after completing the program?

CONTACTS AND LOCATIONS:
Overall Officials: Tatja Hirvikoski, Associate Professor, Principal Investigator — Karolinska Insitutet
Locations (1):
- Habilitering & Hälsa, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Derived] Backman A, Roll-Pettersson L, Mellblom A, Norman-Claesson E, Sundqvist E, Zander E, Vigerland S, Hirvikoski T. Internet-Delivered Psychoeducation (SCOPE) for Transition-Aged Autistic Youth: Pragmatic Randomized Controlled Trial. J Med Internet Res. 2024 Nov 28;26:e49305. doi: 10.2196/49305. PMID 39608000